CLINICAL TRIAL: NCT05657366
Title: The Effect of Peritoneal Lavage on the Incidence of Pancreatic Fistula and Related Complications After Pancreatoduodenectomy in Patients With Different Pancreatic Fistula Risk Scores
Brief Title: Peritoneal Lavage on the Incidence of Pancreatic Fistula and Related Complications After Pancreatoduodenectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: zyeyPDlavage
Record Dates: First submitted 2022-11-07; First posted 2022-12-20 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2022-11

CONDITIONS: Pancreatic Fistula; Pancreaticoduodenal; Fistula
MeSH Terms: conditions — Pancreatic Fistula; Fistula | interventions — Peritoneal Lavage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low and medium risk（a-FRS）lavage (Experimental): alternative pancreatic fistula risk score system，a-FRS Low risk group (0~5%), medium risk group (>5%~20%), lavage
  Interventions: Procedure: Peritoneal lavage
- low and medium risk（a-FRS） no lavage (No Intervention): alternative pancreatic fistula risk score system，a-FRS Low risk group (0~5%), medium risk group (>5%~20%), no lavage
- high risk（a-FRS）lavage (Experimental): alternative pancreatic fistula risk score system，a-FRS high risk group (>20%) lavage
  Interventions: Procedure: Peritoneal lavage
- high risk（a-FRS）no lavage (No Intervention): alternative pancreatic fistula risk score system，a-FRS high risk group (>20%) no lavage

INTERVENTIONS:
Procedure: Peritoneal lavage — Continuous abdominal flushing with normal saline
  Arms: high risk（a-FRS）lavage; low and medium risk（a-FRS）lavage

SUMMARY:
As one of the possible strategies to prevent pancreatic fistula, peritoneal lavage is still widely used in clinical practice, but it lacks more evidence of evidence-based medicine and recommendations of guidelines. Some clinicians believe that routine flushing after pancreatoduodenectomy wastes medical resources and has a negative impact on patients' comfort.

In this study, the investigators designed a multicenter prospective controlled trial to compare the effects of peritoneal lavage and natural drainage on the incidence of pancreatic fistula and related complications after pancreatoduodenectomy. To study the indications of peritoneal lavage.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative diagnosis was pancreatic head, lower common bile duct, ampulla and duodenum tumors;
2. Patients with resectable tumors evaluated by imaging examination, and patients who plan to undergo pancreatoduodenectomy;
3. Subjects informed consent, understood and were willing to cooperate with the trial protocol, and signed relevant documents.

Exclusion Criteria:

1. Complicated with severe liver, kidney, heart, brain, lung and other organ complications;
2. Intraoperative changes in surgical methods, such as patients with tumor dissemination and only abdominal opening and closing; Or it needs to be resected in combination with other organs;
3. Patients and their families do not understand the treatment implementation plan of this study;
4. Failure to complete follow-up;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative Pancreatic Fistula (POPF) | 30 days post-operative
  Presence of Amylase > 3 times the upper limit of normal in surgical drains

SECONDARY OUTCOMES:
Biliary fistula | 90 days post-operative
  Output of bile from drains on or by POD 3, pancreaticojejunostomy leak should be ruled out
Post-Pancreatectomy Hemorrhage | 90 days post-operative
  As defined by the International Study Group for Pancreatic Surgery (ISGPS), grade A, B and C rates
Mortality | 90 days post-operative
  Death related to surgical morbidity
Delayed Gastric Emptying | 90 days post-operative
  As defined by ISGPS, grade A, B and C rates
Abdominal abscess or infection | 90 days post-operative
  Collection >5cm in size, containing gas bubbles, determining systemic signs of infection
Gastrojejunal/Duodenojejunal fistula | 90 days post-operative
  Fistula from gastro/duodenojejunostomy
Wound infection | 90 days post-operative
  Superficial and Deep Surgical Site Incisional Infection
Length of Hospital Stay | 1 year post-operative
  calculated from the day of surgery to the day of discharge, adding up the days after a possible re-admission
Reoperation | 90 days post-operative
  Need for new surgery due to severe morbidity
Readmission | 30 days post-operative
  New admission within 30-days of discharge from hospital
drainage tube duration | 90 days post-operative
  Retention time of abdominal drainage tube

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol